CLINICAL TRIAL: NCT00313105
Title: Smoking Cessation by Nurses With Smokeless Tobacco Buccal Tablets, Nicotine Buccal Tablets, Nicotine Patches With Repeated Therapy Every 6 Months for 2 Years
Brief Title: Smoking Cessation With Smokeless Tobacco, Nicotine Tablets and Nicotine Patches
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University Hospital, Gentofte, Copenhagen (Other)
Collaborators: Danish Research Foundation, FSS, Copenhagen, Denmark (Unknown)
Responsible Party: Philip Tønnesen, M.D., Gentofte Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2005-004626-10
Record Dates: First submitted 2006-04-10; First posted 2006-04-11 (Estimated); Last update posted 2009-09-15 (Estimated); Status verified 2009-09

CONDITIONS: Tobacco Dependence
Keywords: smoking cessation; smokeless tobacco; nicotine patch; nicotine buccal tablets; retreatment; adherence
MeSH Terms: conditions — Tobacco Use Disorder; Smoking Cessation; Tobacco Use | interventions — Tobacco, Smokeless

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Smokeless Tobacco (Experimental): Smokeless Tobacco and individual visits
  Interventions: Drug: Smokeless tobacco (Oliver Twist pellets); Behavioral: smoking cessation counseling
- Nicotine tablets (Active Comparator): Nicotine tablets
  Interventions: Behavioral: smoking cessation counseling
- 3 (Placebo Comparator): 7-mg nicotine patch acts as placebo
  Interventions: Behavioral: smoking cessation counseling

INTERVENTIONS:
Drug: Smokeless tobacco (Oliver Twist pellets) — individual visits with counseling
  Arms: Smokeless Tobacco
Behavioral: smoking cessation counseling — individual visits

SUMMARY:
To test if smokeless tobacco is more effective than nicotine buccal tablets in smoking cessation compared with a control group with low dose nicotine patches.

Also retreatment will be tested with smokeless tobacco every 6 months in failures for 1½ year. Adherence to the program will be enhanced by assessment of cholesterol, blood pressure, lung function and body weight every 6 months for 2 years.

DETAILED DESCRIPTION:
This is an open randomized controlled trial with 3 groups testing smokeless tobacco in smoking cessation: 200 smokers will get smokeless tobacco for 3 months, 200 will get nicotine buccal tablets for 3 months and 200 will get 7-mg nicotine patches for 3 months (control arm). After ½, 1 and 1½ a year failures will get smokeless tobacco in the first 2 groups, while only 7 mg nicotine patches in control group until 1½ year where failures in this group also will get smokeless tobacco. Every ½ year cholesterol, blood pressure, lung function and BMI will be assessed and used to enhance adherence of the participants in this trial.

ELIGIBILITY:
Inclusion Criteria:

* smokers (>7 cig/day)
* Healthy
* Allowed: treated hypertension, diabetes treated with tablets, increased cholesterol,other "mild" diseases
* mild asthma and COPD,
* Motivated to quit smoking
* Motivated to follow the protocol
* Motivated to use medication in this trial

Exclusion Criteria:

* Severe diseases
* Psychiatric diseases
* Used NRT or Zyban the last 2 weeks
* Stopped smoking >2 days during last 3 months
* More than 6 alcoholic drinks per day
* Smokes other products than cigarettes
* Pregnant of lactating

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2006-04; Primary Completion 2010-04 (Estimated); Study Completion 2010-08 (Estimated)

PRIMARY OUTCOMES:
Abstinence from smoking after ½ year (point and continuous abstinence) | 6 months from entry

SECONDARY OUTCOMES:
Adverse events between 3 arms | Up to 6 months from entry
Biomarkers of inhalation between 3 arms (p-cotinine and p-thiocynate and u-NNAL) | 3 and 6 months from entry
Adherence to study | 6,12,24 months from entry
Effect of retreatment (abstinence after 1, 1½ and 2 years) | 12,18 and 24 months from entry
Changes in cholesterol, blood-pressure, lung function, body-weight across smoking status | 6,12,24 months from entry

CONTACTS AND LOCATIONS:
Overall Officials: Philip Tønnesen, M.D., Ph.D., Principal Investigator — Chair dept. pulm. medicine, Gentofte Hospital
Locations (1):
- Dept. pulmonary medicine Y, Gentofte University Hospital, Copenhagen, Hellerup, Denmark